CLINICAL TRIAL: NCT00938964
Title: Lidocaine For Neuroprotection During Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); CAS Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00015641; R01HL096978 (NIH)
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Cognitive Decline
Keywords: Cognition
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Experimental): Lidocaine infusion for 48 hours
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Normal saline infusion for 48 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — Lidocaine versus placebo infusion for 48 hours
  Arms: Lidocaine
Drug: Placebo — Lidocaine versus placebo infusion for 48 hours
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if a drug called lidocaine prevents cognitive injury (a decline in mental abilities) after heart surgery. Lidocaine is currently FDA approved and is commonly used for treating some heart rhythm disorders and for regional anesthesia (blocking nerves). The investigators are enrolling subjects in this research project to see if lidocaine will reduce the high incidence of cognitive injury seen after heart surgery. As part of this study, the investigators will also evaluate the relationship between cognitive injury and genetic makeup and the chemical changes in the subjects blood during and after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. CABG, CABG + Valve, or Valve surgery
2. Use of cardiopulmonary bypass

Exclusion Criteria:

1. Less than 50 years of age
2. History of diabetes
3. History of symptomatic cerebrovascular disease (e.g. prior stroke) with residual deficit
4. Alcoholism (> 2 drinks/day)
5. History of psychiatric illness (any clinical diagnoses requiring therapy)
6. History of drug abuse (any illicit drug use in the past 3 months)
7. Hepatic insufficiency (liver function tests > 1.5 times the upper limit of normal)
8. Severe pulmonary insufficiency (requiring home oxygen therapy)
9. Renal failure (baseline serum creatinine > 2.0 mg/dl)
10. Pregnant women
11. Unable to read and thus unable to complete the cognitive testing
12. Score < 24 on a baseline Mini Mental State examination (MMSE) or greater than or equal to 27 on the baseline Center for Epidemiological Studies Depression (CES-D) Scale -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2016-07-18 (Actual); Study Completion 2017-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Mathew, M. D., Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia

REFERENCES:
- [Background] Newman MF, Kirchner JL, Phillips-Bute B, Gaver V, Grocott H, Jones RH, Mark DB, Reves JG, Blumenthal JA; Neurological Outcome Research Group and the Cardiothoracic Anesthesiology Research Endeavors Investigators. Longitudinal assessment of neurocognitive function after coronary-artery bypass surgery. N Engl J Med. 2001 Feb 8;344(6):395-402. doi: 10.1056/NEJM200102083440601. PMID 11172175
- [Background] Newman MF, Grocott HP, Mathew JP, White WD, Landolfo K, Reves JG, Laskowitz DT, Mark DB, Blumenthal JA; Neurologic Outcome Research Group and the Cardiothoracic Anesthesia Research Endeavors (CARE) Investigators of the Duke Heart Center. Report of the substudy assessing the impact of neurocognitive function on quality of life 5 years after cardiac surgery. Stroke. 2001 Dec 1;32(12):2874-81. doi: 10.1161/hs1201.099803. PMID 11739990
- [Background] Phillips-Bute B, Mathew JP, Blumenthal JA, Grocott HP, Laskowitz DT, Jones RH, Mark DB, Newman MF. Association of neurocognitive function and quality of life 1 year after coronary artery bypass graft (CABG) surgery. Psychosom Med. 2006 May-Jun;68(3):369-75. doi: 10.1097/01.psy.0000221272.77984.e2. PMID 16738066
- [Background] Mathew JP, Mackensen GB, Phillips-Bute B, Grocott HP, Glower DD, Laskowitz DT, Blumenthal JA, Newman MF; Neurologic Outcome Research Group (NORG) of the Duke Heart Center. Randomized, double-blinded, placebo controlled study of neuroprotection with lidocaine in cardiac surgery. Stroke. 2009 Mar;40(3):880-7. doi: 10.1161/STROKEAHA.108.531236. Epub 2009 Jan 22. PMID 19164788
- [Background] Evans DE, Kobrine AI, LeGrys DC, Bradley ME. Protective effect of lidocaine in acute cerebral ischemia induced by air embolism. J Neurosurg. 1984 Feb;60(2):257-63. doi: 10.3171/jns.1984.60.2.0257. PMID 6693953
- [Background] Mitchell SJ. Lidocaine in the treatment of decompression illness: a review of the literature. Undersea Hyperb Med. 2001 Fall;28(3):165-74. PMID 12067153
- [Background] Astrup J, Sorensen PM, Sorensen HR. Inhibition of cerebral oxygen and glucose consumption in the dog by hypothermia, pentobarbital, and lidocaine. Anesthesiology. 1981 Sep;55(3):263-8. doi: 10.1097/00000542-198109000-00013. PMID 7270951
- [Background] Weber ML, Taylor CP. Damage from oxygen and glucose deprivation in hippocampal slices is prevented by tetrodotoxin, lidocaine and phenytoin without blockade of action potentials. Brain Res. 1994 Nov 21;664(1-2):167-77. doi: 10.1016/0006-8993(94)91967-4. PMID 7895026
- [Background] Ayad M, Verity MA, Rubinstein EH. Lidocaine delays cortical ischemic depolarization: relationship to electrophysiologic recovery and neuropathology. J Neurosurg Anesthesiol. 1994 Apr;6(2):98-110. doi: 10.1097/00008506-199404000-00005. PMID 8012179
- [Background] LoPachin RM, Gaughan CL, Lehning EJ, Weber ML, Taylor CP. Effects of ion channel blockade on the distribution of Na, K, Ca and other elements in oxygen-glucose deprived CA1 hippocampal neurons. Neuroscience. 2001;103(4):971-83. doi: 10.1016/s0306-4522(01)00035-5. PMID 11301205
- [Background] Zhang Y, Lipton P. Cytosolic Ca2+ changes during in vitro ischemia in rat hippocampal slices: major roles for glutamate and Na+-dependent Ca2+ release from mitochondria. J Neurosci. 1999 May 1;19(9):3307-15. doi: 10.1523/JNEUROSCI.19-09-03307.1999. PMID 10212290
- [Background] Fujitani T, Adachi N, Miyazaki H, Liu K, Nakamura Y, Kataoka K, Arai T. Lidocaine protects hippocampal neurons against ischemic damage by preventing increase of extracellular excitatory amino acids: a microdialysis study in Mongolian gerbils. Neurosci Lett. 1994 Sep 26;179(1-2):91-4. doi: 10.1016/0304-3940(94)90942-3. PMID 7845632
- [Background] Diaz L, Gomez A, Bustos G. Lidocaine reduces the hypoxia-induced release of an excitatory amino acid analog from rat striatal slices in superfusion. Prog Neuropsychopharmacol Biol Psychiatry. 1995 Sep;19(5):943-53. doi: 10.1016/0278-5846(95)00122-c. PMID 8539430
- [Background] Dutka AJ, Mink R, McDermott J, Clark JB, Hallenbeck JM. Effect of lidocaine on somatosensory evoked response and cerebral blood flow after canine cerebral air embolism. Stroke. 1992 Oct;23(10):1515-20; discussion 1520-1. doi: 10.1161/01.str.23.10.1515. PMID 1412590
- [Background] Evans DE, Kobrine AI. Reduction of experimental intracranial hypertension by lidocaine. Neurosurgery. 1987 Apr;20(4):542-7. doi: 10.1227/00006123-198704000-00006. PMID 3587544
- [Background] Shokunbi MT, Gelb AW, Peerless SJ, Mervart M, Floyd P. An evaluation of the effect of lidocaine in experimental focal cerebral ischemia. Stroke. 1986 Sep-Oct;17(5):962-6. doi: 10.1161/01.str.17.5.962. PMID 3764968
- [Background] Sakabe T, Maekawa T, Ishikawa T, Takeshita H. The effects of lidocaine on canine cerebral metabolism and circulation related to the electroencephalogram. Anesthesiology. 1974 May;40(5):433-41. doi: 10.1097/00000542-197405000-00004. No abstract available. PMID 4822388
- [Background] Johns RA, DiFazio CA, Longnecker DE. Lidocaine constricts or dilates rat arterioles in a dose-dependent manner. Anesthesiology. 1985 Feb;62(2):141-4. doi: 10.1097/00000542-198502000-00008. PMID 3970363
- [Background] Lei B, Popp S, Capuano-Waters C, Cottrell JE, Kass IS. Lidocaine attenuates apoptosis in the ischemic penumbra and reduces infarct size after transient focal cerebral ischemia in rats. Neuroscience. 2004;125(3):691-701. doi: 10.1016/j.neuroscience.2004.02.034. PMID 15099683
- [Background] MacGregor RR, Thorner RE, Wright DM. Lidocaine inhibits granulocyte adherence and prevents granulocyte delivery to inflammatory sites. Blood. 1980 Aug;56(2):203-9. No abstract available. PMID 7397378
- [Background] Schmidt W, Schmidt H, Bauer H, Gebhard MM, Martin E. Influence of lidocaine on endotoxin-induced leukocyte-endothelial cell adhesion and macromolecular leakage in vivo. Anesthesiology. 1997 Sep;87(3):617-24. doi: 10.1097/00000542-199709000-00023. PMID 9316968
- [Background] Lan W, Harmon D, Wang JH, Ghori K, Shorten G, Redmond P. The effect of lidocaine on in vitro neutrophil and endothelial adhesion molecule expression induced by plasma obtained during tourniquet-induced ischaemia and reperfusion. Eur J Anaesthesiol. 2004 Nov;21(11):892-7. doi: 10.1017/s0265021504000249. PMID 15717706
- [Background] Mitchell SJ, Benson M, Vadlamudi L, Miller P. Cerebral arterial gas embolism by helium: an unusual case successfully treated with hyperbaric oxygen and lidocaine. Ann Emerg Med. 2000 Mar;35(3):300-3. doi: 10.1016/s0196-0644(00)70086-2. PMID 10692202
- [Background] Mitchell SJ, Pellett O, Gorman DF. Cerebral protection by lidocaine during cardiac operations. Ann Thorac Surg. 1999 Apr;67(4):1117-24. doi: 10.1016/s0003-4975(99)00057-0. PMID 10320260
- [Background] Wang D, Wu X, Li J, Xiao F, Liu X, Meng M. The effect of lidocaine on early postoperative cognitive dysfunction after coronary artery bypass surgery. Anesth Analg. 2002 Nov;95(5):1134-41, table of contents. doi: 10.1097/00000539-200211000-00002. PMID 12401580
- [Background] Murkin JM, Newman SP, Stump DA, Blumenthal JA. Statement of consensus on assessment of neurobehavioral outcomes after cardiac surgery. Ann Thorac Surg. 1995 May;59(5):1289-95. doi: 10.1016/0003-4975(95)00106-u. No abstract available. PMID 7733754
- [Background] Rey A. L'examen clinique en psychologie. Paper presented at : Presses Universitaires de France, 1964; Paris
- [Background] Randt C, Brown E. Administration Manual: Randt Memory Test. New Youk Life Sciences Associates; 1983
- [Background] Wechsler D. The Wechsler Adult Intelligence Sacle-Revised (Manual): Psychological Corporation: 1981.
- [Background] Reitan RM. Validity of the trail making test as an indicator of organic brain damage. Percept Mot Skills, 1958; 8:271-276
- [Background] Ruff RM, Parker SB. Gender- and age-specific changes in motor speed and eye-hand coordination in adults: normative values for the Finger Tapping and Grooved Pegboard Tests. Percept Mot Skills. 1993 Jun;76(3 Pt 2):1219-30. doi: 10.2466/pms.1993.76.3c.1219. PMID 8337069
- [Background] Murkin JM, Stump DA, Blumenthal JA, McKhann G. Defining dysfunction: group means versus incidence analysis--a statement of consensus. Ann Thorac Surg. 1997 Sep;64(3):904-5. doi: 10.1016/s0003-4975(97)00743-1. No abstract available. PMID 9307516
- [Background] Lyden P, Brott T, Tilley B, Welch KM, Mascha EJ, Levine S, Haley EC, Grotta J, Marler J. Improved reliability of the NIH Stroke Scale using video training. NINDS TPA Stroke Study Group. Stroke. 1994 Nov;25(11):2220-6. doi: 10.1161/01.str.25.11.2220. PMID 7974549
- [Background] Roach GW, Newman MF, Murkin JM, Martzke J, Ruskin A, Li J, Guo A, Wisniewski A, Mangano DT. Ineffectiveness of burst suppression therapy in mitigating perioperative cerebrovascular dysfunction. Multicenter Study of Perioperative Ischemia (McSPI) Research Group. Anesthesiology. 1999 May;90(5):1255-64. doi: 10.1097/00000542-199905000-00006. PMID 10319770
- [Background] Mark DB, Nelson C, Delong E, et al. Comparisin of quality of life outcomes following coronary angioplasty, coronary bypass surgery and medicine. J Am Coll Cardiol. 1993; 21:216A
- [Background] Cleary PD, Greenfield S, McNeil BJ. Assessing quality of life after surgery. Control Clin Trials. 1991 Aug;12(4 Suppl):189S-203S. doi: 10.1016/s0197-2456(05)80023-6. PMID 1663855
- [Background] Hlatky MA, Boineau RE, Higginbotham MB, Lee KL, Mark DB, Califf RM, Cobb FR, Pryor DB. A brief self-administered questionnaire to determine functional capacity (the Duke Activity Status Index). Am J Cardiol. 1989 Sep 15;64(10):651-4. doi: 10.1016/0002-9149(89)90496-7. PMID 2782256
- [Background] Ware JE Jr. Standards for validating health measures: definition and content. J Chronic Dis. 1987;40(6):473-80. doi: 10.1016/0021-9681(87)90003-8. PMID 3298292
- [Background] Guyatt GH, Sullivan MJ, Thompson PJ, Fallen EL, Pugsley SO, Taylor DW, Berman LB. The 6-minute walk: a new measure of exercise capacity in patients with chronic heart failure. Can Med Assoc J. 1985 Apr 15;132(8):919-23. PMID 3978515
- [Background] Goldman L, Hashimoto B, Cook EF, Loscalzo A. Comparative reproducibility and validity of systems for assessing cardiovascular functional class: advantages of a new specific activity scale. Circulation. 1981 Dec;64(6):1227-34. doi: 10.1161/01.cir.64.6.1227. PMID 7296795
- [Background] McDowell I, Newell C. Measuring Health: A Guide To Rating Scales And Questionnaires. New York: Oxford University Press; 1987.
- [Background] Bergner M, Bobbitt RA, Carter WB, Gilson BS. The Sickness Impact Profile: development and final revision of a health status measure. Med Care. 1981 Aug;19(8):787-805. doi: 10.1097/00005650-198108000-00001. PMID 7278416
- [Background] Wassertheil-Smoller S, Blaufox MD, Oberman A, Davis BR, Swencionis C, Knerr MO, Hawkins CM, Langford HG. Effect of antihypertensives on sexual function and quality of life: the TAIM Study. Ann Intern Med. 1991 Apr 15;114(8):613-20. doi: 10.7326/0003-4819-114-8-613. PMID 2003706
- [Background] Cronbach LJ. Essentials of Psycological Testing. New York: Harper and Row; 1970
- [Background] Benjamini Y, Hochberg Y. Controlling the False Discovery Rate: A Practical and Powerful Approach to Multiple Testing. J R Statist Soc B. 1995;57(1):289-300
- [Derived] Klinger RY, Cooter M, Berger M, Podgoreanu MV, Stafford-Smith M, Ortel TL, Welsby IJ, Levy JH, Rinder HM, Newman MF, Mathew JP; Neurologic Outcomes Research Group (NORG) of The Duke Heart Center. Effect of intravenous lidocaine on the transcerebral inflammatory response during cardiac surgery: a randomized-controlled trial. Can J Anaesth. 2016 Nov;63(11):1223-32. doi: 10.1007/s12630-016-0704-0. Epub 2016 Jul 28. PMID 27470233

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 550 participants consented; 478 participants were randomized.
Period: Overall Study
Arm/Group | Lidocaine | Placebo
Started | 241 | 237
Completed | 211 | 209
Not Completed | 30 | 28
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 22 | 18
Not completed — Found to Meet Exclusion Criteria | 3 | 4

BASELINE CHARACTERISTICS:
Population: Number of participants who completed the study are included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Placebo | Total
Number analyzed (Participants) | 211 | 209 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (9.1) | 66.5 (9.5) | 66.7 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 49 | 109
  Male | 151 | 160 | 311
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 211 | 209 | 420

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function From Baseline Characterized as Continuous Cognitive Change
Description: To characterize cognitive function over time, while minimizing potential redundancy in the cognitive measures, a factor analysis was performed on the 14 cognitive test scores from baseline. We chose a five-factor solution, which represents 5 cognitive domains: structured verbal memory, unstructured verbal memory, executive function, visual memory and attention/concentration. To quantify overall cognitive function, a baseline cognitive index was first calculated as the mean of the 5 preoperative domain scores. The cognitive index score has a mean of zero, thus any positive score is above the mean, any negative score is below the mean. A continuous change score was then calculated by subtracting the baseline from the 6-week cognitive index. The resulting outcome measure is unbounded with standard deviation of 0.35. A negative change score indicating decline and a positive score indicating improvement.
Time Frame: Preoperative to 6 weeks after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 211 | 209
units on a scale | 0.07 (0.32) | 0.07 (0.37)

2. Primary Outcome: Count of Participants With a Decline of Greater Than or Equal to One Standard Deviation in One or More of Five Cognitive Domain Scores Reported as a Dichotomous Post-operative Cognitive Deficit (POCD) Outcome
Description: To characterize cognitive function over time, while minimizing potential redundancy in the cognitive measures, a factor analysis was performed on the 14 cognitive test scores from baseline. We chose a five-factor solution, which represents 5 cognitive domains: structured verbal memory, unstructured verbal memory, executive function, visual memory and attention/concentration. Each domain score is normally distributed with a mean of zero. A change score was calculated for each domain by subtracting the baseline from the 6-week score. A dichotomous outcome variable of post-operative cognitive deficit was defined as a decline of ≥1 standard deviation in 1 or more of the 5 domains.
Time Frame: Preoperative to 6 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 211 | 209
Participants | 87 | 83

3. Secondary Outcome: Transcerebral Activation Gradients of Platelets
Description: Paired jugular venous and radial arterial blood samples were drawn at baseline, cross-clamp removal, end of cardiopulmonary bypass, and 6 hours post cross-clamp removalime points and analyzed by fluorescence-activated cell sorting to identify activated platelets. Transcerebral activation gradients were calculated by subtracting arterial values from venous values and were compared between groups
Time Frame: Baseline to 6 hours post cross-clamp removal
Population: Planned substudy, that was analyzed after 202 enrolled subjects
Measure: Mean (Standard Deviation); unit: Mean linear fluorescence intensity-MLFI
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 105 | 97
Mean linear fluorescence intensity-MLFI
  Baseline | -0.03 (0.79) | 0.35 (1.91)
  Cross-clamp removal | 0.03 (1.21) | 0.43 (1.44)
  End of Bypass | 0.33 (3.25) | 0.05 (2.65)
  6 hours post cross-clamp removal | 0.37 (2.65) | 0.27 (1.07)

4. Secondary Outcome: Transcerebral Activation Gradients of Neutrophils
Description: Paired jugular venous and radial arterial blood samples were drawn at baseline, cross-clamp removal, end of cardiopulmonary bypass, and 6 hours post cross-clamp removal and analyzed by fluorescence-activated cell sorting to identify activated platelets. Transcerebral activation gradients were calculated by subtracting arterial values from venous values and were compared between groups
Time Frame: Baseline to 6 hours post cross-clamp removal
Population: Planned substudy, that was analyzed after 202 enrolled subjects
Measure: Mean (Standard Deviation); unit: Mean linear fluorescence intensity-MLFI
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 105 | 97
Mean linear fluorescence intensity-MLFI
  Baseline | -2.02 (8.15) | -0.08 (9.17)
  Cross-clamp removal | 0.56 (6.82) | 0.17 (5.53)
  End of Bypass | 0.58 (4.54) | 1.19 (6.76)
  6 hours post cross-clamp removal | 1.04 (7.08) | -0.68 (8.61)

5. Secondary Outcome: Transcerebral Activation Gradients of Monocytes
Description: as for outcome 3
Time Frame: Baseline to 6 hours post cross-clamp removal
Population: Planned substudy, that was analyzed after 202 enrolled subjects.
Measure: Mean (Standard Deviation); unit: Mean linear fluorescence intensity-MLFI
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 105 | 97
Mean linear fluorescence intensity-MLFI
  Baseline | -4.22 (19.10) | -0.04 (17.78)
  Cross-clamp removal | -2.46 (16.94) | 1.83 (16.80)
  End of Bypass | -0.34 (19.57) | 2.64 (15.69)
  6 hours post cross-clamp removal | 1.21 (15.08) | 0.54 (13.69)

6. Secondary Outcome: Transcerebral Activation Gradient of Platelet-neutrophil Conjugates
Description: as for outcome 3
Time Frame: Baseline to 6 hours post cross-clamp removal
Population: Planned substudy, that was analyzed after 202 enrolled subjects.
Measure: Mean (Standard Deviation); unit: Mean linear fluorescence intensity-MLFI
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 105 | 97
Mean linear fluorescence intensity-MLFI
  Baseline | -0.15 (9.64) | -0.43 (8.40)
  Cross-clamp removal | 0.02 (4.33) | -0.73 (3.97)
  End of Bypass | -0.73 (4.99) | -0.40 (5.12)
  6 hours post cross-clamp removal | -0.10 (5.40) | 0.19 (4.73)

7. Secondary Outcome: Change in Cognitive Function From Baseline
Description: To characterize cognitive function over time, while minimizing potential redundancy in the cognitive measures, a factor analysis was performed on the 14 cognitive test scores from baseline. We chose a five-factor solution, which represents 5 cognitive domains: structured verbal memory, unstructured verbal memory, executive function, visual memory and attention/concentration. To quantify overall cognitive function, a baseline cognitive index was first calculated as the mean of the 5 preoperative domain scores. The cognitive index score has a mean of zero, thus any positive score is above the mean, any negative score is below the mean. A continuous change score was then calculated by subtracting the baseline from the 1 year cognitive index. The resulting outcome measure is unbounded with standard deviation of 0.35. A negative change score indicating decline and a positive score indicating improvement
Time Frame: 1 year after surgery
Population: There was 26 lidocaine patients and 17 placebo patients lost to follow-up between the primary 6-week follow-up and the final 1-year follow-up time point. Only those returning for 1 year follow-up were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 185 | 192
units on a scale | 0.09 (0.34) | 0.07 (0.34)

8. Secondary Outcome: Change in Duke Activity Status Index (DASI)
Description: The DASI is a 12-item scale of functional capacity that has been found to correlate well with objective measures of maximal exercise capacity. Items reflect activities of personal care, ambulation, household tasks, sexual function, and recreational activities. Activities done "with no difficulty" receive scores, which are weighted and summed, for a quantitative measure of functional status. Scores range from 0 to 60; a higher-weighted score indicates better function.
Time Frame: baseline, 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 211 | 209
units on a scale | -10.98 (15.4) | -11.67 (16.8)

9. Secondary Outcome: Change in Duke Activity Status Index (DASI)
Description: as for outcome 8
Time Frame: baseline, 1-year
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 185 | 192
units on a scale | 6.3 (18.3) | 6.96 (16.9)

10. Secondary Outcome: Change in Neurological Function, as Measured by the National Institutes of Health Stroke Scale (NIHSS)
Description: The National Institutes of Health Stroke Scale (NIHSS) is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The range of scores is from 0 (normal) to 42 (profound effect of stroke on patient).
Time Frame: baseline, 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 211 | 209
units on a scale | 0.05 (0.5) | 0.04 (0.5)

11. Secondary Outcome: Change in Neurological Function, as Measured by the National Institutes of Health Stroke Scale (NIHSS)
Description: as for outcome 10
Time Frame: baseline, 1-year
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 185 | 192
units on a scale | 0.05 (0.70) | 0.07 (0.60)

12. Secondary Outcome: Change in Center for Epidemiological Studies Depression Scale (CES-D)
Description: Center for Epidemiological Studies Depression Scale (CES-D). The CES-D is a 20-item self-report examination designed to measure symptoms of depression. Subjects rate the degree to which they have experienced a range of symptoms of depression, such as "I had crying spells" and "I felt lonely." Scores range from 0 to 60, with higher scores indicating greater depressive symptoms. Scores greater than 16 are typically considered indicative of clinically significant depression.
Time Frame: baseline, 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 211 | 209
units on a scale | 0.57 (7.5) | 0.16 (8.3)

13. Secondary Outcome: Change in Center for Epidemiological Studies Depression Scale (CES-D)
Description: as for outcome 12
Time Frame: baseline, 1-year
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 185 | 192
units on a scale | -1.27 (7.7) | -0.89 (7.9)

14. Secondary Outcome: Change in Spielberger State Anxiety Inventory (STAI)
Description: Spielberger State Anxiety Inventory (STAI): The STAI consists of two 20-item scales that measure anxiety. Representative items include statements such as "I feel nervous" and "I feel worried." These items are rated on a 4-point scale, based on how well they describe the patient's current or typical mood, from "not at all" to "very much so." Scores range from 20 to 80, with higher scores indicating greater anxiety.
Time Frame: baseline, 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 211 | 209
units on a scale | -7.12 (12.1) | -6.31 (11.4)

15. Secondary Outcome: Change in Spielberger State Anxiety Inventory (STAI)
Description: as for outcome 14
Time Frame: baseline, 1-year
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 185 | 192
units on a scale | -6.70 (12.7) | -6.39 (10.3)

16. Secondary Outcome: Change in Symptom Limitations
Description: Symptom limitations: Patients were given a list of eight symptoms and asked to rate the degree to which the symptom limited daily activities. The symptoms were angina, shortness of breath, arthritis, back trouble, leg pains, headaches, fatigue, and other. Scores range from 8 to 32, with higher scores indicating greater limitations.
Time Frame: baseline, 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 211 | 209
units on a scale | -0.67 (4.0) | -0.8 (3.9)

17. Secondary Outcome: Change in Symptom Limitations
Description: as for outcome 16
Time Frame: baseline, 1-year
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 185 | 192
units on a scale | -1.39 (3.8) | -1.48 (3.8)

18. Secondary Outcome: Change in the Duke Older Americans Resources and Services Procedures- Instrumental Activities of Daily Living (OARS-IADL)
Description: Duke Older Americans Resources and Services Procedures- Instrumental Activities of Daily Living (OARS-IADL): This measure contains six items that assess the ability to perform important tasks for daily living (e.g., "Could you prepare your own meals?" "Could you drive a car?"). Scores range from 6 to 24. Higher scores indicate increasing difficulty in engaging in daily activities.
Time Frame: baseline, 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 211 | 209
units on a scale | 2.46 (4.2) | 2.1 (3.9)

19. Secondary Outcome: Change in the Duke Older Americans Resources and Services Procedures- Instrumental Activities of Daily Living (OARS-IADL)
Description: as for outcome 18
Time Frame: baseline, 1-year
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 185 | 192
units on a scale | -0.15 (2.1) | -0.31 (2.6)

20. Secondary Outcome: Change in the Cognitive Difficulties Scale
Description: Cognitive Difficulties Scale: a 39-item scale, is a self-report assessment of perceived problems in long- and short-term memory, concentration, attention, and psycho-motor coordination. Sample items are "I forget errands I planned to do" and "I fail to recognize people I know." Scores range from 39 to 164, with higher scores indicating greater cognitive difficulty.
Time Frame: baseline, 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 211 | 209
units on a scale | -3 (14.6) | -3.21 (15.9)

21. Secondary Outcome: Change in the Cognitive Difficulties Scale
Description: as for outcome 20
Time Frame: baseline, 1-year
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 185 | 192
units on a scale | -0.46 (16.1) | -1.02 (17)

22. Secondary Outcome: Change in Perceived Social Support
Description: Perceived Social Support Scale: Twelve items indicate how strongly subjects agree that there is "a special person who is around when I am in need" and "my family really tries to help me." Choices range from "very strongly disagree" to "very strongly agree." Items are summed for a range of 12 to 84, with a high score meaning more social support.
Time Frame: baseline, 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 211 | 209
units on a scale | 1.23 (14) | -0.49 (13.9)

23. Secondary Outcome: Change in Perceived Social Support
Description: as for outcome 22
Time Frame: baseline, 1-year
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 185 | 192
units on a scale | 0.71 (13.4) | -1.16 (12.9)

24. Secondary Outcome: Change in Social Activity
Description: Social Activity: This measure consisted of eight items that indicate the degree of social interaction. Sample items are "How often do you talk on the telephone with friends and relatives?" and "How often do you attend meetings of social groups, clubs, or civic organizations?" Scores range from 8 to 32. A lower score indicates more social activity.
Time Frame: baseline, 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 211 | 209
units on a scale | 0.95 (3.4) | 1.59 (3.2)

25. Secondary Outcome: Change in Social Activity
Description: as for outcome 24
Time Frame: baseline, 1-year
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 185 | 192
units on a scale | -0.20 (3.2) | 0.03 (3.4)

26. Secondary Outcome: Change in Study 36-Item Short Form Health Survey (SF-36)
Description: The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36): The SF-36 was designed to measure general health status. Two scales were used: Work Activities (four items) and General Health (one item). For the work activities scale, the reported score was the sum of four questions, each with values ranging from 1 to 4, the total score could range from 4 to 16. A higher score on Work Activities indicates more health-related problems For the general health question, the patients ranked their health from Excellent (1) to poor (5), the scale ranged from 1 to 5 with 1 being best health and 5 being worst. A high score in General Health indicates poorer health state.
Time Frame: baseline, 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 211 | 209
units on a scale
  6-Week Change Work activities | 2.71 (4.9) | 3 (4.3)
  6-Week Change General health perception | -0.004 (1.3) | -0.03 (1.2)

27. Secondary Outcome: Change in Study 36-Item Short Form Health Survey (SF-36)
Description: as for outcome 26
Time Frame: baseline, 1-year
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 185 | 192
units on a scale
  1 year Change Work Activities | -1.37 (4.3) | -1.42 (4.1)
  1 year Change General health perception | -0.28 (1.2) | -0.43 (1.1)

28. Secondary Outcome: Change in Neurological Function, as Measured by the Western Perioperative Neurologic Scale (WPNS)
Description: The Western perioperative neurologic scale was designed to detect neurologic deficits after cardiac surgery. It includes 14 items classified into eight domains (mentation, speech, cranial nerve function, motor weakness, sensation and cerebellum, reflexes, and gait). Each item is scored from 0 (severe deficit) to3 (normal), and a maximum score of 42 indicates normal neurological function.
Time Frame: baseline, 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 211 | 209
units on a scale | 0.04 (1.10) | -0.01 (1.3)

29. Secondary Outcome: Change in Neurological Function, as Measured by the Western Perioperative Neurologic Scale (WPNS)
Description: as for outcome 28
Time Frame: baseline, 1-year
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 185 | 192
units on a scale | 0.02 (1.10) | -0.02 (1.20)

ADVERSE EVENTS:
Time Frame: Adverse events were collected until hospital discharge (approximately 4 -10 days) . Serious Adverse Events were reported up to one year.
Arm/Group | Lidocaine | Placebo
All-Cause Mortality (participants affected / at risk) | 6/241 | 7/237
Serious Adverse Events (participants affected / at risk) | 105/241 | 103/237
Other Adverse Events (participants affected / at risk) | 34/241 | 34/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine (N=241) | Placebo (N=237)
Acute Blood Loss anemia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Acute Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 6 (6)
Anaphylatic or Anaphylactoid rxn (Immune system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Atrial Dysrhythmia - Atrial Fibrillation (Cardiac disorders) | 41 (41) | 41 (41)
Atrial Dysrhythmia -Sinus Bradycardia (Cardiac disorders) | 0 (0) | 4 (4)
AV Block (Cardiac disorders) | 1 (1) | 1 (1)
Bacermia/sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bleeding (Blood and lymphatic system disorders) | 6 (6) | 7 (7)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 4 (4)
Chylothorax (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Complete heart block (Cardiac disorders) | 7 (7) | 6 (6)
Confusion/encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 2 (2) | 0 (0)
Continuous coma (Nervous system disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Diaphragmic tear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dysphagia (Nervous system disorders) | 1 (1) | 1 (1)
Fever of Non-Specified Origin (Immune system disorders) | 0 (0) | 1 (1)
Fluid overload (General disorders) | 1 (1) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 2 (2) | 0 (0)
Heart attack-hospitalization (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemorrhagic shock (Cardiac disorders) | 2 (2) | 0 (0)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemophilus Influenzae (Infections and infestations) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 6 (6) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypotension (Cardiac disorders) | 8 (8) | 7 (7)
Hypothermia (Nervous system disorders) | 0 (0) | 1 (1)
Hypovolemic shock (Cardiac disorders) | 1 (1) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 6 (6)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Junctional rhythm (Cardiac disorders) | 5 (5) | 3 (3)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Left brachial embolectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Left bundle branch block (Cardiac disorders) | 0 (0) | 1 (1)
Left pleural effusion thoracentesis (Surgical and medical procedures) | 0 (0) | 1 (1)
Left vocal cord palsy (Nervous system disorders) | 0 (0) | 1 (1)
Leukocytosis (Infections and infestations) | 8 (8) | 7 (7)
LVAD (Surgical and medical procedures) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MRSA (Infections and infestations) | 2 (2) | 0 (0)
Nausea/Vomiting/Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4)
Pacemaker Placement (Surgical and medical procedures) | 6 (6) | 8 (8)
Pain (General disorders) | 1 (1) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
PEA Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 3 (3)
Phlebitis (Immune system disorders) | 1 (1) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Prolonged hospitalization (General disorders) | 1 (1) | 0 (0)
Protein malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (2)
re-admission after fall (General disorders) | 2 (2) | 0 (0)
Reexploration For Bleeding (Surgical and medical procedures) | 4 (4) | 4 (4)
Reintubation (Surgical and medical procedures) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 7 (7) | 5 (5)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Shock (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 2 (2)
Sternal Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Stroke (Vascular disorders) | 2 (2) | 6 (6)
Subcutaneous Air (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Suprapubic catheter placement (Surgical and medical procedures) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Thoracentesis (Surgical and medical procedures) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8) | 8 (8)
Thrush (Infections and infestations) | 0 (0) | 1 (1)
Tranfusion rxn (Immune system disorders) | 0 (0) | 1 (1)
Trifascicular block (Cardiac disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 3 (3) | 1 (1)
Ventilation > 48hr (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ventilator associated pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Ventricular Dysrhythmia - Ventricular Tachycardia (Cardiac disorders) | 2 (2) | 5 (5)
Ventricular ectopy (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine (N=241) | Placebo (N=237)
Atrial Dysrhythmia - Atrial Fibrillation (Cardiac disorders) | 34 (34) | 34 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No